CLINICAL TRIAL: NCT04187014
Title: Oral Tranexamic Acid vs. Oral Aminocaproic Acid to Reduce Blood Loss, Transfusion Index and Complications After Total Hip Replacement. A Prospective, Randomized, Double Blind Clinical Trial
Brief Title: Oral Tranexamic Acid vs. Oral Aminocaproic Acid to Reduce Blood Loss After Total Hip Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carlos A Acosta-Olivo (Other)
Responsible Party: Sponsor-Investigator, Carlos A Acosta-Olivo, Professor, Universidad Autonoma de Nuevo Leon
Organization: Universidad Autonoma de Nuevo Leon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OR19-00003
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Blood Loss, Surgical
Keywords: Total hip replacement; Oral tranexamic acid; Oral aminocaproic acid; Blood loss
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — Aminocaproic Acid; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Two study groups will be generated, each consisting of 45 research subjects, randomly each recipient will receive 3 doses of one of the two study drugs (tranexamic acid or aminocaproic acid). The group to which the patient belongs will be assigned through a computer program, the patient will not know to which group he belongs or what medication he will receive. The patients will be extracted from the external traumatology clinic
Who Masked: Participant, Investigator
Masking Description: Prior to being included in the study, the patient will be mentioned the times when he will receive the medication as well as the dosage of administration. The patient will not know what medication is being administered to him / her. The pills will be given to the patient in a medicine cup without access to any information legend. In the same way, the medication will be administered by a doctor outside the research protocol and will not participate in any other phase of the study so that no member of the research team will know what medication was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (Active Comparator): Will be administered orally three times (administering 2 tablets each time). In the case of tranexamic acid are 650 mg each. The first administration will be two hours before the induction of anesthesia, the second 6 hours post-surgery and the third 12 hours after surgery. All by oral administration with a drink of water. The medicines will be administered with a volume of 40 ml of water.
  For tranexamic acid a total dose of 3.9 grams (6 tablets) divided between the 3 administrations (1.3 grams each, ie 2 tablets of 650 mg) will be administered.
  Interventions: Drug: Tranexamic acid tablets
- Aminocaproic acid (Experimental): Will be administered orally three times (administering 2 tablets each time). In the case of aminocaproic tablets are 1000 mg each.The first administration will be two hours before the induction of anesthesia, the second 6 hours post-surgery and the third 12 hours after surgery. All by oral administration with a drink of water. The medicines will be administered with a volume of 40 ml of water.
  For the aminocaproic acid, a total dose of 6 grams (6 tablets) divided between the 3 administrations (2 gram each, ie 2 tablets of 1000 mg) will be administered.
  Interventions: Drug: Aminocaproic Acid 1000Mg Tab

INTERVENTIONS:
Drug: Aminocaproic Acid 1000Mg Tab — Oral administration of a total 6 g of aminocaproic acid to reduce blood loss
  Other Names: Oral administration of aminocaproic acid
  Arms: Aminocaproic acid
Drug: Tranexamic acid tablets — Oral administration of 3.9 g of tranexamic acid to reduce blood loss
  Other Names: Oral administration of tranexamic acid
  Arms: Tranexamic acid

SUMMARY:
This study compares two oral medications (tranexamic acid and aminocaproic acid) as hemostatic agent administered in patients undergoing primary total hip replacement

DETAILED DESCRIPTION:
With the aging population, the incidence of joint osteoarthritis is rising. Total hip arthroplasty (THA) is one of the most common surgeries used for the treatment of end-stage degenerative hip disease, which is almost always accompanied by joint pain, deformity and motor dysfunction.

Few articles have compared TXA and ε-ACA in joint arthroplasties. Whether ε-ACA has comparable hemostatic effects compared with TXA is unknown. A recent systematic review compared the effectiveness of TXA versus ε-ACA administered intravenously as a hemostatic agent in patients who had undergone a TKA and THR, and the results showed that the total blood loss was greater in the ε-ACA groups, but no significant differences between the two groups regarding transfusion rates were identified (Liu et al., 2018).

Regarding oral administration, two clinical trials compared the use of oral TXA versus intravenous and topical in patients who had undergone THA, reaching the conclusion that if efficiency, safety, and cost are considered the main crucial parameters during the evaluation of TXA administration methods, oral TXA stands as an efficacious, safe, and low-cost method to reduce blood loss after THA compared with the IV and topical forms. Additionally, considering the ease of drug administration in the tablet form, oral TXA appears to represent a superior mode of administration than IV and topical TXA (Kayupov et al., 2017; Luo et al., 2018).

The investigator's work team previously published a randomized controlled clinical trial in which it prospectively compared blood loss, transfusion rate and complications similar to this study but in total primary knee replacement, finding no differences with respect to any of the parameters studied except for the adverse effects, which were greater for the group that received tranexamic acid, this study was the first to compare the oral administration of these two medications in the field of orthopedics (Morales-Avalos et al., 2019) and the present protocol wants to do it now in the total primary hip replacement which is well known to be associated with greater blood loss than total knee replacement.

HYPOTHESIS: There are no significant differences in blood loss (total blood loss, external blood loss, hidden blood loss, intraoperative blood loss and drainage output), transfusion index, complications and hemoglobin/hematocrit levels in patients undergoing total hip prostheses treated with tranexamic acid or aminocaproic acid orally.

General objectives To compare the effect of oral aminocaproic acid as a hemostatic agent against oral tranexamic acid administered preoperatively and postoperatively in patients undergoing elective surgery of total hip replacement.

Specific objectives

1. Selection and randomization of patients.
2. Performing total hip replacement surgery and administration of AAC or AXA according to randomization and the methodology established in this protocol
3. Establishment of a protocol for the administration of aminocaproic acid orally for its use as a hemostatic agent in elective surgery of total hip replacement.
4. Determination of total blood loss, external blood loss, hidden blood loss, transfusion index, decrease in hemoglobin/hematocrit levels, drainage volume, intrahospital stay, analogous visual scale and SF-12 scale between tranexamic acid and the aminocaproic acid, both orally, in each group in the pre-operatively, trans operatively and post-operatively established times and compare them statistically.
5. Determine and record the possible complications and side effects observed with the use of both drugs included in the study.
6. Determine the cost and monetary savings associated with the administration of each drug.
7. Comparison and statistical analysis of the results between the study groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Total replacement of the primary hip due to: 1) Primary Coxarthrosis, 2) Avascular hip necrosis, 3) Transcervical fracture
3. Unilateral procedure
4. Press-fit prosthesis
5. Without the use of cement for the placement of the prosthesis
6. Desire to participate voluntarily in the study and signature of informed consent
7. Pre-operative assessment with result between ASA I, ASA II or ASA III performed and annexed in the clinical file either by the Department of Internal Medicine, Cardiology or Anesthesiology of our hospital.
8. Possibility for oral administration of the drug.

Exclusion Criteria:

1. History of thrombotic or embolic event in the last 6 months
2. Clinical history of coagulopathy
3. Previous surgeries in the hip to intervene
4. Patients who have received aspirin, platelet or coumarinic antiplatelet agents in the week prior to surgery or NSAIDs two days prior to surgery.
5. History of myocardial infarction, arteriopathy or unstable angina in the 12 months prior to surgery.
6. Those patients whose preoperative assessment corresponds to an ASA IV or the procedure is contraindicated in its preoperative assessment.
7. Revision hip replacement
8. Tumoral hip replacement
9. Bilateral hip replacement
10. Cognitive deficit
11. Patients who meet the inclusion criteria but do not wish to participate in the study
12. Patients with a diagnosis of Terminal Chronic Kidney Disease or with a serum creatinine higher than 1.47 mg / dl in the preoperative laboratories.
13. Patients with inability to ingest the drug orally.
14. Patients who are pregnant or breast-feeding or who are taking oral contraceptives.
15. Seizure history
16. Hypersensitivity to the active substance or to any of the excipients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Total blood loss (TBL) | The third day postoperative,at the time of obtaining the result of the hematocrit of 72 hours
  Total blood loss 72 hours after surgery,The Gross and Nadler formula was used to calculate TBL. TBL = patient's blood volume (PBV) x (Hctpre - Hctpost)/Hctave (Hctpre = the initial pre-operative Hct level, Hctpost = the Hct on the morning of POD3). PBV = k1 x height (m) + k2 x weight (kg) + k3 (k1 = 0.3669, k2 = 0.03219, and k3 = 0.6041 for men; and k1 = 0.3561, k2 = 0.03308, and k3 = 0.1833 for women, Hctave = the average of the Hctpre and Hctpost)
External blood loss (EBL) | On the second postoperative day (48 hours), when removing the surgical drainage.]
  External blood loss (EBL) was estimated by adding the intraoperative bleeding and the blood in the drain collectors upon removal after 48 hours
Hidden blood loss (HBL) | The third day postoperative
  Defined as total blood loss minus external blood loss

SECONDARY OUTCOMES:
Change in hematocrit level | Hematocrit levels will be measured at 24, 48 and 72 hours postsurgery
  Hematocrit levels obtained in 3 samples taken at different times postsurgery
Drainage quantification | Drainage quantification will be registered at 24 and 48 hours postsurgery
  Drainage will be quantified in ml at 2 different times postsurgery
Therapeutic effect on visual analog scale | Pain will be measured at 24, 48 and 72 hours postsurgery
  The Visual Analog Scale is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (scale of 10). It will be assessed as a numeric scale from 0 to 10.
Change in Hemoglobin level | Hemoglobin levels will be measured at 24, 48 and 72 hours postsurgery
  Hemoglobin levels will be obtained in 3 samples taken at different times postsurgery
Rate of complications | at 24, 48 and 72 hours, 7 days, 4 and 6 weeks
  Complications related to the surgery or to the administration of the study medication
Rate of transfusion | at 24, 48 and 72 hours, 7 days, 4 and 6 weeks
  Need to administer globular packages following the indications of transfusion haemoglobin (Hb) of 8 g/dl in patients free of cardiovascular disease and Hb of 9 g/dl in patients with established cardiovascular disease or cardiovascular risk factors with symptoms of anaemia (defined as bad mental status, palpitation, or shortness of breath not due to other causes). Hb below 10 g/dl in patients with poor clinical tolerance of lower values was also an indication for transfusion. Symptoms of poor clinical tolerance of lower values were signs of hypoxia such as tachycardia, dyspnoea or syncope or drainage of more than 1 l of blood in the first 24 hours
Rate of intraoperative blood loss | Immediately after the end of the surgery
  Intra-operative blood loss was calculated using the difference between the weights of the used gauze and the original unused gauze (25 cm x 25 cm, monolayer, weight of 30 grams), in addition to the blood volume accumulated in suction bottles subtracting the volume of saline solution during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, PhD, Study Chair — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kayupov E, Fillingham YA, Okroj K, Plummer DR, Moric M, Gerlinger TL, Della Valle CJ. Oral and Intravenous Tranexamic Acid Are Equivalent at Reducing Blood Loss Following Total Hip Arthroplasty: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Mar 1;99(5):373-378. doi: 10.2106/JBJS.16.00188. PMID 28244907
- [Result] Luo ZY, Wang HY, Wang D, Zhou K, Pei FX, Zhou ZK. Oral vs Intravenous vs Topical Tranexamic Acid in Primary Hip Arthroplasty: A Prospective, Randomized, Double-Blind, Controlled Study. J Arthroplasty. 2018 Mar;33(3):786-793. doi: 10.1016/j.arth.2017.09.062. Epub 2017 Oct 6. PMID 29107495
- [Result] Liu Q, Geng P, Shi L, Wang Q, Wang P. Tranexamic acid versus aminocaproic acid for blood management after total knee and total hip arthroplasty: A systematic review and meta-analysis. Int J Surg. 2018 Jun;54(Pt A):105-112. doi: 10.1016/j.ijsu.2018.04.042. Epub 2018 May 1. PMID 29723672
- [Result] Morales-Avalos R, Ramos-Morales T, Espinoza-Galindo AM, Garay-Mendoza D, Pena-Martinez VM, Marfil-Rivera LJ, Garza-Ocanas L, Acosta-Olivo C, Cerda-Barbosa JK, Valdes-Gonzalez NL, Vilchez-Cavazos F. First Comparative Study of the Effectiveness of the Use of Tranexamic Acid against epsilon-Aminocaproic Acid via the Oral Route for the Reduction of Postoperative Bleeding in TKA: A Clinical Trial. J Knee Surg. 2021 Mar;34(4):383-405. doi: 10.1055/s-0039-1696722. Epub 2019 Sep 6. PMID 31491796